CLINICAL TRIAL: NCT00379470
Title: A Prospective, Multi-center Trial of NovoTTF-100A Compared to Best Standard of Care in Patients With Progressive or Recurrent GBM
Brief Title: Effect of NovoTTF-100A in Recurrent Glioblastoma Multiforme (GBM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF-11
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Recurrent Glioblastoma Multiforme
Keywords: Brain tumor; Treatment; Minimal toxicity; GBM; Glioblastoma; Recurrent; TTFields
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Best Standard of Care (Active Comparator): Patients randomized to the BSC group will be treated with one chemotherapy according to the BSC practiced at each center.
  Interventions: Device: NovoTTF-100A
- NovoTTF-100A (Experimental)
  Interventions: Device: NovoTTF-100A

INTERVENTIONS:
Device: NovoTTF-100A — multiple four-week courses of continuous NovoTTF-100A treatment

SUMMARY:
The study is a randomized, controlled trial, designed to test the efficacy and safety of a new medical device, the NovoTTF-100A. The device is an experimental, portable, battery operated device for chronic treatment of patients with recurrent or progressive glioblastoma multiforme (GBM) using alternating electric fields (termed TTFields).

DETAILED DESCRIPTION:
PAST CLINICAL EXPERIENCE:

The effect of the electric fields generated by the NovoTTF-100A device (TTFields) has been tested in two pilot trials in humans. The data from these trials suggest NovoTTF-100A may improve time to disease progression and overall survival of recurrent GBM patients. Although the number of patients in the pilot trials is small, The FDA has determined that the data gathered so far warrant testing of NovoTTF-100A treatment as a possible therapy for patients with recurrent GBM.

DESCRIPTION OF THE TRIAL:

Patients with GBM whose disease has recurred or progressed despite standard treatment (Surgery, radiation therapy, Temozolomide treatment) and meet all of the requirements for participation in the study will be randomly assigned to one of two groups:

1. Treatment with the NovoTTF-100A device, or
2. Treatment with the best standard of care practiced at each of the participating centers.

If assigned to the best standard of care group, patients will receive a chemotherapeutic agent chosen based on their prior treatments and the standard of care practiced at each treating center.

If assigned to the NovoTTF-100A group, the patients will be treated continuously for as long as their disease is stable or regressing. NovoTTF-100A treatment will consist of wearing four electrically insulated electrodes on the head. Electrode placement will require shaving of the scalp before treatment. After an initial short hospitalization (24 hours) patients will be released to continue treatment at home where they can maintain their regular daily routine.

During the trial, regardless of whether assigned to the NovoTTF-100A treatment group or the best standard of care group, patients will need to return once every month the hospital outpatient clinics where they will be examined by a physician and undergo routine laboratory examinations. These routine visits will continue for as long as the patient's disease is not progressing. After progression, if such occurs, patients will need to return once per month for two more months to the outpatient clinic for similar follow up examinations.

During the visits to the clinic patients will be examined physically and neurologically. Additionally, routine blood tests and ECG will be performed. A routine MRI of the head will be performed at baseline and after 2, 4 and 6 months. After this follow up plan, patients will be contacted once per month by telephone to answer basic questions about their health status.

SCIENTIFIC BACKGROUND:

Electric fields exert forces on electric charges similar to the way a magnet exerts forces on metallic particles within a magnetic field. These forces cause movement and rotation of electrically charged biological building blocks, much like the alignment of metallic particles seen along the lines of force radiating outwards from a magnet.

Electric fields can also cause muscles to twitch and if strong enough may heat tissues. TTFields are alternating electric fields of low intensity. This means that they change their direction repetitively many times a second. Since they change direction very rapidly (200 thousand times a second), they do not cause muscles to twitch, nor do they have any effects on other electrically activated tissues in the body (brain, nerves and heart). Since the intensities of TTFields in the body are very low, they do not cause heating.

The breakthrough finding made by NovoCure was that finely tuned alternating fields of very low intensity, now termed TTFields (Tumor Treating Fields), cause a significant slowing in the growth of cancer cells. Due to the unique geometric shape of cancer cells when they are multiplying, TTFields cause the building blocks of these cells to move and pile up in such a way that the cells physically explode. In addition, cancer cells also contain miniature building blocks which act as tiny motors in moving essential parts of the cells from place to place. TTFields cause these tiny motors to fall apart since they have a special type of electric charge.

As a result of these two effects, cancer tumor growth is slowed and can even reverse after continuous exposure to TTFields.

Other cells in the body (normal healthy tissues) are affected much less than cancer cells since they multiply at a much slower rate if at all. In addition TTFields can be directed to a certain part of the body, leaving sensitive areas out of their reach.

In conclusion, TTField hold the promise of serving as a brand new cancer treatment with very few side effects and promising affectivity in slowing or reversing this disease.

ELIGIBILITY:
Inclusion Criteria:

* Pathological evidence of GBM using WHO classification criteria.
* > 18 years of age.
* Not a candidate for further radiotherapy or additional resection of residual tumor.
* Patients with disease progression (by Macdonald criteria i.e., > 25% or new lesion) documented by CT or MRI within 4 weeks prior to enrollment
* Karnofsky scale ≥ 70
* Life expectancy at least 3 months
* Participants of childbearing age must use effective contraception.
* All patients must sign written informed consent.

Exclusion Criteria:

* Actively participating in another clinical treatment trial
* Within 4 weeks from surgery for recurrence
* Within 4 weeks from any prior chemotherapy.
* Within 4 weeks from radiation therapy
* Pregnant
* Significant co-morbidities (within 4 weeks prior to enrollment):

  1. Significant liver function impairment - AST or ALT > 3 times the upper limit of normal
  2. Total bilirubin > upper limit of normal
  3. Significant renal impairment (serum creatinine > 1.7 mg/dL)
  4. Coagulopathy (as evidenced by PT or APTT >1.5 times control in patients not undergoing anticoagulation)
  5. Thrombocytopenia (platelet count < 100 x 103/μL)
  6. Neutropenia (absolute neutrophil count < 1 x 103/μL)
  7. Anemia (Hb < 10 g/L)
  8. Severe acute infection
* Implanted pacemaker, defibrillator or deep brain stimulator, or documented clinically significant arrhythmias.
* Infra-tentorial tumor
* Evidence of increased intracranial pressure (midline shift > 5mm, clinically significant papilledema, vomiting and nausea or reduced level of consciousness)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2006-09; Primary Completion 2009-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 2 years from initiation of accrual

SECONDARY OUTCOMES:
Progression free survival at 6 months (PFS6) | 2 years from initiation of accrual
Median Time to Disease Progression (TTP) | 2 years from initiation of accrual
% 1-year survival | 2 years from initiation of accrual
Radiological response (Macdonald criteria) | 2 years from initiation of accrual
Quality of life assessment (EORTC QLQ-C30) | 2 years from initiation of accrual
Adverse events severity and frequency | 2 years from initiation of accrual

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Gutin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Roger Stupp, MD, Principal Investigator — University of Lausanne Hospital - Multidisciplinary Oncology Center
Locations (25):
- United States (15):
  - Northwestern University, Chicago, Illinois
  - University of Illinois in Chicago, Chicago, Illinois
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Boston University Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - NJ Neuroscience Institute - JFK Medical Center, Edison, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Columbia University Medical Center, New York, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- University Hospital Graz, Graz, Austria
- Czechia (2):
  - FN Brno - Masaryk University, Brno
  - Na Homolce Hospital, Prague
- France (2):
  - Hospital of Neurology Lyon - University Claude Bernard Lyon 1, Lyon
  - Group Hospitals Pitie-Salpetriere, Paris
- Germany (3):
  - University Hospital Augsburg, Augsburg
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - University Hospital of Schleswig-Holstein, Kiel
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

REFERENCES:
- [Background] Kirson ED, Gurvich Z, Schneiderman R, Dekel E, Itzhaki A, Wasserman Y, Schatzberger R, Palti Y. Disruption of cancer cell replication by alternating electric fields. Cancer Res. 2004 May 1;64(9):3288-95. doi: 10.1158/0008-5472.can-04-0083. PMID 15126372
- [Background] Kirson ED, Dbaly V, Tovarys F, Vymazal J, Soustiel JF, Itzhaki A, Mordechovich D, Steinberg-Shapira S, Gurvich Z, Schneiderman R, Wasserman Y, Salzberg M, Ryffel B, Goldsher D, Dekel E, Palti Y. Alternating electric fields arrest cell proliferation in animal tumor models and human brain tumors. Proc Natl Acad Sci U S A. 2007 Jun 12;104(24):10152-7. doi: 10.1073/pnas.0702916104. Epub 2007 Jun 5. PMID 17551011
- [Background] Salzberg M, Kirson E, Palti Y, Rochlitz C. A pilot study with very low-intensity, intermediate-frequency electric fields in patients with locally advanced and/or metastatic solid tumors. Onkologie. 2008 Jul;31(7):362-5. doi: 10.1159/000137713. Epub 2008 Jun 24. PMID 18596382
- [Derived] Stupp R, Wong ET, Kanner AA, Steinberg D, Engelhard H, Heidecke V, Kirson ED, Taillibert S, Liebermann F, Dbaly V, Ram Z, Villano JL, Rainov N, Weinberg U, Schiff D, Kunschner L, Raizer J, Honnorat J, Sloan A, Malkin M, Landolfi JC, Payer F, Mehdorn M, Weil RJ, Pannullo SC, Westphal M, Smrcka M, Chin L, Kostron H, Hofer S, Bruce J, Cosgrove R, Paleologous N, Palti Y, Gutin PH. NovoTTF-100A versus physician's choice chemotherapy in recurrent glioblastoma: a randomised phase III trial of a novel treatment modality. Eur J Cancer. 2012 Sep;48(14):2192-202. doi: 10.1016/j.ejca.2012.04.011. Epub 2012 May 18. PMID 22608262